CLINICAL TRIAL: NCT02904915
Title: Paracervical Block Versus No Paracervical Block During IUD Insertion
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Pamela Berens, Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-16-0664
Record Dates: First submitted 2016-09-08; First posted 2016-09-19 (Estimated); Results first posted 2018-11-07 (Actual); Last update posted 2018-11-07 (Actual); Status verified 2018-10

CONDITIONS: Analgesia; IUD Insertion
MeSH Terms: conditions — Agnosia | interventions — Lidocaine; Intrauterine Devices

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Paracervical block (Active Comparator): Intrauterine device (IUD) placement with paracervical block with 1% lidocaine.
  Interventions: Drug: Lidocaine; Device: Intrauterine device (IUD)
- No analgesia (Active Comparator): IUD placement with no analgesia.
  Interventions: Other: No analgesia; Device: Intrauterine device (IUD)

INTERVENTIONS:
Drug: Lidocaine — Intrauterine device (IUD) placement with paracervical block with 1% lidocaine.
  Other Names: xylocaine, lignocaine
  Arms: Paracervical block
Other: No analgesia — IUD placement without analgesia.
  Arms: No analgesia
Device: Intrauterine device (IUD) — IUD placement with or without paracervical block with 1% lidocaine.

SUMMARY:
The purpose of this study is to compare the pain level and level of discomfort with paracervical block versus no analgesia in women who present to the University of Texas (UT) Physicians Obstetrics and Gynecology Continuity Clinic, The UT Physicians Women's Center, and the UT Physicians Women's Center- Bellaire for IUD insertion.

ELIGIBILITY:
Inclusion Criteria:

* Women of reproductive age who present for an IUD insertion procedure at the University of Texas Physicians Obstetrics and Gynecology Continuity Clinic, The UT Physicians Women's Center, and the UT Physicians Women's Center- Bellaire for IUD insertion.

Exclusion Criteria:

* Women with current pelvic inflammatory disease (PID)
* Women who are not good candidates for an IUD
* Patients who have a Lidocaine allergy

Ages: 18 Years to 52 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2017-01-12 (Actual); Primary Completion 2017-10-09 (Actual); Study Completion 2017-10-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pamela D Berens, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Paracervical Block | No Analgesia
Started | 25 | 25
Completed | 25 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Paracervical Block | No Analgesia | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.6 (4.6) | 26.6 (5.9) | 25.6 (5.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 25 | 50
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 12 | 14 | 26
  Caucasian | 3 | 3 | 6
  Hispanic | 7 | 7 | 14
  Asian | 1 | 0 | 1
  Unknown | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 25 | 25 | 50
Prior delivery type [Count of Participants; unit: Participants]
  Cesarean Section | 7 | 4 | 11
  Vaginal | 15 | 21 | 36
  None | 3 | 0 | 3
Contraception History [Count of Participants; unit: Participants]
  Oral contraceptive pill | 6 | 2 | 8
  Intrauterine device (IUD) | 1 | 5 | 6
  Nexplanon/injectables | 1 | 0 | 1
  Depo Provera/injections | 7 | 3 | 10
  Condoms (female and male) | 3 | 2 | 5
  Nuvaring | 1 | 6 | 7
  None | 3 | 4 | 7
  Unknown | 3 | 3 | 6
History of Infection [Count of Participants; unit: Participants]
  Chlamydia | 0 | 2 | 2
  Bacterial vaginosis (BV) | 8 | 13 | 21
  Yeast | 4 | 3 | 7
  Human papillomavirus (HPV) | 6 | 4 | 10
  None | 7 | 3 | 10
Take pain medication [Count of Participants; unit: Participants] | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Pain Score as Assessed by a Visual Analogue Scale (VAS)
Description: The order of overall events are: insertion of speculum, assessment of pain via a visual analogue scale (VAS) (about 30 seconds after insertion of the speculum), injection of 2cc 1% lidocaine at the tenaculum site of the cervix, placement of tenaculum (about 2-3 minutes after insertion of speculum), assessment of pain via VAS (about 30 seconds after insertion of the tenaculum), injection of 3cc 1% lidocaine at the 4 and 8 o'clock position of the cervix, insert IUD (about 4-5 minutes after insertion of tenaculum), and assessment of pain via VAS (about 30 seconds after insertion of the IUD).
  The Faces pain VAS was used, which ranges from 0 (very happy, no hurt) to 10 (hurts as much as you can imagine).
Time Frame: baseline (about 30 seconds after insertion of the speculum)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Paracervical Block | No Analgesia
Number analyzed (Participants) | 25 | 25
units on a scale | 2.4 (2.3) | 2.1 (2.4)
Statistical Analysis 1: Comparison: Paracervical Block vs No Analgesia; Test type: Superiority; p = 0.59, Fisher Exact

2. Primary Outcome: Pain Score as Assessed by a Visual Analogue Scale
Description: as for outcome 1
Time Frame: about 30 seconds after insertion of the tenaculum (tenaculum inserted about 2 to 3 minutes after insertion of speculum)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Paracervical Block | No Analgesia
Number analyzed (Participants) | 25 | 25
units on a scale | 2.1 (2.5) | 2.7 (2.4)
Statistical Analysis 1: Comparison: Paracervical Block vs No Analgesia; Test type: Superiority; p = 0.39, Fisher Exact

3. Primary Outcome: Pain Score as Assessed by a Visual Analogue Scale
Description: as for outcome 1
Time Frame: about 30 seconds after insertion of the IUD (IUD inserted about 4 to 5 minutes after insertion of tenaculum)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Paracervical Block | No Analgesia
Number analyzed (Participants) | 25 | 25
units on a scale | 2.6 (2.7) | 3.6 (2.9)
Statistical Analysis 1: Comparison: Paracervical Block vs No Analgesia; Test type: Superiority; p = 0.23, Fisher Exact

ADVERSE EVENTS:
Time Frame: From time of speculum placement until the patient left the office (patient leaves office about 3-5 minutes after the procedure, for a total of about 15 minutes from speculum placement to leaving the office).
Arm/Group | Paracervical Block | No Analgesia
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25

LIMITATIONS AND CAVEATS:
No Sham Block. Subjects had more variability in baseline pain scores (taken after speculum placement but prior to any procedure) than anticipated, and thus the study was underpowered.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-04): https://cdn.clinicaltrials.gov/large-docs/15/NCT02904915/Prot_SAP_000.pdf